CLINICAL TRIAL: NCT02750943
Title: A Clinical Study Investigating the Gingivitis Efficacy of a Stannous Fluoride Dentifrice
Brief Title: Potential of Stannous Fluoride Toothpaste to Reduce Gum Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205045
Record Dates: First submitted 2015-11-02; First posted 2016-04-26 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stannous Fluoride (Experimental): Participants will apply a full ribbon of dentifrice containing 0.454% w/w stannous fluoride to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening)
  Interventions: Drug: Stannous Fluoride
- Sodium Monofluorophosphate (Active Comparator): Participants will apply a full ribbon of dentifrice containing Dentifrice containing 1000ppm fluoride as sodium monofluorophosphate to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening)
  Interventions: Drug: Sodium Monofluorophosphate

INTERVENTIONS:
Drug: Stannous Fluoride — Dentifrice containing 0.454% w/w stannous fluoride
  Arms: Stannous Fluoride
Drug: Sodium Monofluorophosphate — Dentifrice containing 1000ppm fluoride as sodium monofluorophosphate
  Arms: Sodium Monofluorophosphate

SUMMARY:
This will be a single-center, 12 week, examiner-blind, randomized, stratified (gender and baseline mean whole mouth MGI score), two-treatment, parallel group, clinical study in healthy adult volunteers with moderate gingivitis. This study will evaluate the efficacy of a dentifrice containing 0.454% weight by weight (w/w) stannous fluoride to control gingivitis and gingival bleeding following 12 weeks twice daily brushing, compared to a negative control dentifrice.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral/dental examination.
* Absence of any condition that would impact on the subject's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* A minimum of 20 permanent gradable teeth. (Gradable teeth are those where restorative materials cover less than 25% of the tooth surface graded).
* Moderate gingivitis present at the screening visit in the opinion of the investigator from a gross visual gingival assessment.
* Visible blood in toothpaste expectorant at Screening and Baseline (Visit 2).

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family.
* An employee of any toothpaste manufacturer or their immediate family.
* Medical History/Current Medication A. Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any other medical condition (e.g. Diabetes Mellitus) that would make the subject unlikely to fully complete the study or any that increases the risk to the subject or undermines the data validity B.Screening i. Currently taking antibiotics or requiring antibiotic use prior to dental prophylaxis or other dental procedures.

ii. Currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.

iii. Currently taking a systemic medication which, in the opinion of the C. Baseline, Day 28 and Day 96 Assessment Visits i. Has taken antibiotics in the previous 14 days. ii. Has taken an anti-inflammatory medication which, in the opinion of the investigator, could affect gingival condition in the previous 14 days.

iii. Has taken a systemic medication which, in the opinion of the investigator, could affect gingival condition in the previous 14 days (e.g. calcium channel blockers, or aspirin therapy).could affect gingival condition in the previous 14 days (e.g. calcium channel blockers, or aspirin therapy).Investigator, could affect gingival condition (e.g. calcium channel blockers, or aspirin therapy).

* Have current active caries or periodontitis that may, in the opinion of the investigator, compromise the study or the oral health of the subjects if they participate in the study.
* Restorations in a poor state of repair.
* Partial dentures or orthodontic appliances.
* Teeth bleaching within 12 weeks of screening.
* Use of a chlorhexidine mouthwash within 14 days of baseline.
* Current smokers or smokers who have quit within the past 6 months prior to screening or subjects currently using smokeless forms of tobacco, e.g. Gutkha, Pan containing tobacco, Pan Masala or nicotine based e-cigarettes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-11-01; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in a single center in Germany.
Pre-assignment Details: A total of 317 participants were screened. Out of which only 253 participants were randomized.
Groups:
- Stannous Fluoride: Participants were instructed to apply a full ribbon of dentifrice containing 0.454% weight by weight (w/w) stannous fluoride to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) for 12 weeks.
- Sodium Monofluorophosphate: Participants were instructed to apply a full ribbon of dentifrice containing 1000 parts per million (ppm) fluoride as sodium monofluorophosphate to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) for 12 weeks.
Period: Overall Study
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Started | 125 | 128
Completed | 119 | 119
Not Completed | 6 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Stannous Fluoride: Participants were instructed to apply a full ribbon of dentifrice containing 0.454% w/w stannous fluoride to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) for 12 weeks.
- Sodium Monofluorophosphate: Participants were instructed to apply a full ribbon of dentifrice containing 1000 ppm fluoride as sodium monofluorophosphate to the study toothbrush and brush their teeth in their usual manner for one timed minute twice daily (morning and evening) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate | Total
Number analyzed (Participants) | 125 | 128 | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.39 (13.610) | 36.37 (13.179) | 37.86 (13.453)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Sites at Week 12
Description: Number of bleeding sites was measured as bleeding index (BI) via a single examiner using a color coded periodontal probe. The probe was engaged approximately 1 millimetre (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI was assessed on the facial and lingual gingival surfaces of each scorable tooth (7-7 in each arch). The BI scoring system used to measure bleeding sites is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. Bleeding sites were assessed as the number of bleeding sites with a BI score of 1 or 2.
Time Frame: Week 12
Population: Intent to treat (ITT) population which included all participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement. Number of participants analyzed is the number of participants from ITT population evaluated for this outcome at Week 12 for respective treatment arm.
Measure: Least Squares Mean (Standard Error); unit: number of bleeding sites
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 119 | 119
number of bleeding sites | 42.02 (1.91) | 67.36 (1.91)
Statistical Analysis 1: Comparison: Stannous Fluoride vs Sodium Monofluorophosphate; Test type: Superiority or Other; p < 0.0001, ANCOVA — From ANCOVA analysis with treatment group, gender and baseline MGI stratification as factors baseline as covariates; Least square (LS) mean difference = -25.340, 95% CI 2-sided [-30.682 to -19.998] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

2. Secondary Outcome: Number of Bleeding Sites at Week 4
Description: Number of bleeding sites was measured as BI via a single examiner using a color coded periodontal probe. The probe was engaged approximately 1 mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI was assessed on the facial and lingual gingival surfaces of each scorable tooth (7-7 in each arch). The BI scoring system used to measure bleeding sites is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed. Bleeding sites were assessed as the number of bleeding sites with a BI score of 1 or 2.
Time Frame: Week 4
Population: Intent to treat (ITT) population which included all participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement. Number of participants analyzed is the number of participants from ITT population evaluated for this outcome at Week 4 for respective treatment arm.
Measure: Least Squares Mean (Standard Error); unit: number of bleeding sites
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 121 | 122
number of bleeding sites | 45.44 (1.92) | 68.30 (1.91)

3. Secondary Outcome: Bleeding Index (BI) at Week 4 and Week 12
Description: BI was assessed by a single examiner using a color coded periodontal probe. The probe was engaged approximately 1mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system to be used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed
Time Frame: Week 4, Week 12
Population: Intent to treat (ITT) population which included all participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement. Number of participants analyzed is the number of participants from ITT population evaluated for this outcome at specific time points for respective treatment arm.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 122 | 123
score on a scale
  BI at Week 4 (n=121, 122) | 0.29 (0.01) | 0.44 (0.01)
  BI at Week 12 (n=119, 119) | 0.27 (0.01) | 0.43 (0.01)

4. Secondary Outcome: Modified Gingival Index (MGI) at Week 4 and Week 12
Description: MGI was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin). The scoring of the MGI was performed under dental office conditions using a standard dental light for illuminating the oral cavity. This procedure was performed by a single examiner. The MGI scoring system is as follows: 0 = absence of inflammation; 1 = mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit; 2 = mild inflammation; criteria as above but involving the entire marginal or papillar gingival units; 3= moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit; 4 = severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.
Time Frame: Week 4, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 122 | 123
score on a scale
  MGI at Week 4 | 2.27 (0.01) | 2.40 (0.01)
  MGI at Week 12 | 2.29 (0.01) | 2.47 (0.01)

5. Secondary Outcome: Number of Participants With Visible Blood in Expectorate (Presence [Trace, Substantial]/Absence) at Week4 and Week 12
Description: Visible blood in expectorate for each participant was classified as (i) Present (Trace or Substantial) (ii) Absent. The number of participants with blood 'Present' (Trace or Substantial) or 'absent' in expectorate was analyzed.
Time Frame: Week 4, Week 12
Population: as for outcome 3
Measure: Number; unit: number of participants
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 122 | 123
number of participants
  At Week 4, Visible blood= Present | 92 | 89
  At Week 4, Visible blood= Trace | 35 | 31
  At Week 4, Visible blood= Substantial | 57 | 58
  At Week 4, Visible blood= Absent | 30 | 34
  At Week 12, Visible blood= Present | 72 | 78
  At Week 12, Visible blood= Trace | 18 | 13
  At Week 12, Visible blood= Substantial | 54 | 65
  At Week 12, Visible blood= Absent | 47 | 41

ADVERSE EVENTS:
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/128
Other Adverse Events (participants affected / at risk) | 20/125 | 22/128
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stannous Fluoride (N=125) | Sodium Monofluorophosphate (N=128)
Oral hyperkeratosis (Gastrointestinal disorders) | 15 | 19
Gingival pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 1
Gingival injury (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.